CLINICAL TRIAL: NCT01890707
Title: A Comparison of the Effect of Intravenous Sedation Versus General Anesthesia in Patients Undergoing Minor Gynecologic Surgery
Brief Title: Intravenous Sedation Versus General Anesthesia in Patients Undergoing Minor Gynecologic Surgery
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Change in procedure.
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Shireen Ahmad, Principal Investigator, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: STU00062431
Record Dates: First submitted 2012-06-01; First posted 2013-07-02 (Estimated); Results first posted 2020-01-02 (Actual); Last update posted 2020-01-02 (Actual); Status verified 2019-12

CONDITIONS: Surgery; Anesthesia; Pain
Keywords: Gynecology; Pain; Anesthesia; Quality of Recovery 40
MeSH Terms: conditions — Pain | interventions — Anesthesia, General; Deep Sedation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Deep Sedation (Active Comparator): Deep sedation
  Interventions: Procedure: Deep Sedation
- General Anesthesia (Other): Administration of general anesthesia. Propofol given IV, succinylcholine and rocuronium given IV and Sevoflurane via the endotracheal tube.
  Interventions: Procedure: General Anesthesia

INTERVENTIONS:
Procedure: General Anesthesia — Administer: Fentanyl:1mcg/kg prior to induction, additional doses to maintain blood pressure and heart rate within 20% of preoperative values, Propofol:2mg/kg,succinylcholine, 0.5mg/kg,to be followed with Rocuronium if necessary,bolus: 0.4mg/kg, Sevoflurane and oxygen to be titrated to maintain BIS value of 40-60.
  Arms: General Anesthesia
Procedure: Deep Sedation — IV administration of Propofol,initial rate 100ug/kg/min, titrated to maintain BIS 65-75,Fentanyl,Ketamine,1mcg/kg,0.5mg/kg,additional 10mg increments for analgesia/movement.
  Arms: Deep Sedation

SUMMARY:
The use of deep sedation may improve the quality of recovery of patients undergoing minor gynecologic procedures. These patients may also have shorter hospital stays and potentially lower healthcare costs. Additionally, the use of deep sedation for second trimester pregnancy termination may be associated with less bleeding, a smaller decrease in perioperative hemoglobin and better quality of recovery.

DETAILED DESCRIPTION:
Once consent for the study has been obtained subjects will be randomly allocated into 2 groups, using a computer generated table of random numbers. Anesthetic management will be standardized (Appendix 1, 2). Group A (study group) will receive deep sedation . Group B (control group) will receive general anesthesia. Subjects will be instructed preoperatively, on the proper use of the verbal rating scale (VRS) for pain and nausea scores. All patients routinely have a blood count checked preoperatively and based on the results are either screened for cross matched for potential transfusion. All subjects will complete the POMS questionnaire preoperatively.

Gestational size will be determined by the surgeon preoperatively using the most recent ultrasound measurements.

Participants will undergo a standard pre-operative evaluation, laboratory testing and laminaria insertion one day prior to surgery in the Family Planning and Contraception Clinic. All subjects will receive a prescription for ibuprofen 600mg and hydrocodone/acetaminophen 5/325mg with standardized instructions to take the last oral dose no later than six hours before the operative time. The last dose medication and time of administration will be recorded.

Intraoperative management:

A standardized intraoperative anesthetic protocol will be utilized by the anesthesia personnel (Appendix #1, 2).Clinical management of excessive intraoperative bleeding will be at the discretion of the anesthesiologist.

Intraoperative red blood cell loss will be estimated based on hematacrit of the contents of suction canister. The surgical field will be draped carefully so that all blood lost will either be collected in the suction canister or the pocket of the vaginal drape, so that it can also be suction into the canister prior to obtaining the laboratory sample. Every attempt will be made by the surgeons to keep all unaccounted blood loss to gloves, instruments, drapes, surgery table and OR floor, to a minimum. The suction tubing will be rinsed with50 mls of saline at the end of the procedure.

All participants will receive a standard paracervical block of 20ml. of 1% lidocaine with 5 units of vasopressin. Further uterotonics or surgical intervention for excessive bleeding will be at the discretion of the surgeon and documented in study data sheets.

Postoperative management:

Immediately postoperatively the surgeon of record will be asked to rate the quality of the anesthesia provided to the patient. He / she will complete a Surgeon Satisfaction with Intraoperative Sedation survey. (Appendix # 3)

In the recovery room, VRS for pain will be assessed upon admission and at 30 minute intervals thereafter. Analgesics will be administered according to the severity of the pain. Subjects will receive oral analgesics unless they are unable to take oral analgesics, in which case IV hydromorphone will be administered.

Vomiting and retching episodes will be assessed at 30 minute intervals using a VRS, and patients with scores greater than 4 or those who request antiemetic treatment will be treated with ondansetron 4mg IV.

Postoperative blood loss will be measured by weighing the patient dressings with a precision computerized scale system prior to discarding them. Prior to the subjects discharge from the facility, a drop of venous blood will be obtained from the existing intravenous catheter, for measurement hemoglobin. Hemoglobin determination of less than 8 gms/dL, will be verified with the hospital laboratory. Management decisions will be made in conjunction with the surgeon, based on the subject's clinical status.

Recovery from anesthesia and return of psychomotor ability will be assessed using the Modified Post Anesthesia Discharge Scoring System (MPADSS, see Appendix #6). A score of > 9 will indicate discharge readiness. Discharge readiness requires that a patient be awake and alert with stable vital signs, able to ambulate without assistance, and free of side effects.

Times from end of surgery to oral intake and readiness for discharge, and all adverse events and medications administered will be recorded. Subjects will be contacted by telephone 24 hours after surgery to obtain post-discharge data, including a QoR-40 assessment and a Pittsburgh Sleep Quality Index survey (PSQI).

Discharge analgesia and antiemetic medications will be standardized.

ELIGIBILITY:
Inclusion Criteria:

* Female patients undergoing second trimester abortions:
* Pregnancy: 12-24 weeks gestational size
* ASA PS I and II
* No history of diabetes mellitus, GERD or sleep apnea
* Age: > 18 years of age
* Fluent in English

Exclusion Criteria:

* ASA PSIII, Emergency surgery
* Pregnancy: > 24 weeks gestational size
* Age: < 18 years of age
* Diabetes mellitus
* Gastroesophageal reflux disease
* Hiatal hernia
* Obstructive sleep apnea
* Coagulopathy
* Chronic pain syndromes
* Chronic opioid dependency
* Alcohol or illicit drug abuse
* BMI: > 35Kg/m2
* Allergy to study protocol drugs

Drop out criteria:

* Subjects withdrawal of consent.
* Subjects who experience massive bleeding intraoperatively, will be excluded from the final data analysis

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2012-10-19 (Actual); Primary Completion 2014-04-15 (Actual); Study Completion 2014-04-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shireen Ahmad, M.D., Principal Investigator — Northwestern University
Locations (1):
- Prentice Womens' Hospital, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sa Rego MM, White PF. What is new in monitored anesthesia care? Curr Opin Anaesthesiol. 1998 Dec;11(6):601-6. doi: 10.1097/00001503-199811000-00003. PMID 17013278
- [Background] Sa Rego MM, Watcha MF, White PF. The changing role of monitored anesthesia care in the ambulatory setting. Anesth Analg. 1997 Nov;85(5):1020-36. doi: 10.1097/00000539-199711000-00012. No abstract available. PMID 9356094
- [Background] Song D, Greilich NB, White PF, Watcha MF, Tongier WK. Recovery profiles and costs of anesthesia for outpatient unilateral inguinal herniorrhaphy. Anesth Analg. 2000 Oct;91(4):876-81. doi: 10.1097/00000539-200010000-00020. PMID 11004041
- [Background] Snyder SK, Roberson CR, Cummings CC, Rajab MH. Local Anesthesia With Monitored Anesthesia Care vs General Anesthesia in Thyroidectomy: A Randomized Study. Arch Surg. 2006 Feb;141(2):167-73. doi: 10.1001/archsurg.141.2.167. PMID 16490894
- [Background] Scarborough DA, Herron JB, Khan A, Bisaccia E. Experience with more than 5,000 cases in which monitored anesthesia care was used for liposuction surgery. Aesthetic Plast Surg. 2003 Nov-Dec;27(6):474-80. doi: 10.1007/s00266-003-3043-9. Epub 2004 Mar 4. PMID 14994165
- [Background] Eldor L, Weissman A, Fodor L, Carmi N, Ullmann Y. Breast augmentation under general anesthesia versus monitored anesthesia care: a retrospective comparative study. Ann Plast Surg. 2008 Sep;61(3):243-6. doi: 10.1097/SAP.0b013e31815bfe98. PMID 18724120
- [Background] EDWARDS G, MORTON HJ, PASK EA, WYLIE WD. Deaths associated with anaesthesia; a report on 1,000 cases. Anaesthesia. 1956 Jul;11(3):194-220. doi: 10.1111/j.1365-2044.1956.tb07975.x. No abstract available. PMID 13340197
- [Background] Warner MA, Shields SE, Chute CG. Major morbidity and mortality within 1 month of ambulatory surgery and anesthesia. JAMA. 1993 Sep 22-29;270(12):1437-41. doi: 10.1001/jama.270.12.1437. PMID 8371443
- [Background] Aldrete JA, Kroulik D. A postanesthetic recovery score. Anesth Analg. 1970 Nov-Dec;49(6):924-34. No abstract available. PMID 5534693
- [Background] White PF. Criteria for fast-tracking outpatients after ambulatory surgery. J Clin Anesth. 1999 Feb;11(1):78-9. doi: 10.1016/s0952-8180(98)00119-6. No abstract available. PMID 10396724
- [Background] Chung F, Chan VW, Ong D. A post-anesthetic discharge scoring system for home readiness after ambulatory surgery. J Clin Anesth. 1995 Sep;7(6):500-6. doi: 10.1016/0952-8180(95)00130-a. PMID 8534468
- [Background] Wong J, Tong D, De Silva Y, Abrishami A, Chung F. Development of the functional recovery index for ambulatory surgery and anesthesia. Anesthesiology. 2009 Mar;110(3):596-602. doi: 10.1097/ALN.0b013e318197a16d. PMID 19212260

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects will be recruited up to 14 days prior to surgery, by either the anesthesiology or the gynecology investigators. A preoperative anesthetic assessment will be completed. Once consent for the study has been obtained subjects will be randomly allocated into 2 groups, using a computer generated table of random numbers.
Period: Overall Study
Arm/Group | Deep Sedation | General Anesthesia
Started | 11 | 8
Completed | 10 | 7
Not Completed | 1 | 1
Not completed — Lost to Follow-up | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Deep Sedation | General Anesthesia | Total
Number analyzed (Participants) | 10 | 7 | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 07 | 17
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 34.3 (3.46) | 35 (7.3) | 34.5 (5.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 7 | 17
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 10 | 7 | 17
Height Inches [Mean (Standard Deviation); unit: Inches] | 67.1 (2.3) | 64 (1.85) | 65.8 (2.16)
Kilogram Weight [Mean (Standard Deviation); unit: Kilogram Weight] | 73.9 (13.8) | 64.6 (6.3) | 70.07 (12.23)
Gestational Age [Median (Standard Deviation); unit: Weeks] | 19.17 (2.13) | 19.85 (2.58) | 19.45 (2.35)

OUTCOME MEASURES:

1. Primary Outcome: Quality of Recovery - 40 Scores
Description: The patients self reported quality of recovery - 40 scores as completed 24 hours after the surgical procedure.
  40 questions regarding the recovery of patients on a 1 poor-5 excellent scale. Total score on scale 40 (poor recovery)-200 (excellent recovery)
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Deep Sedation | General Anesthesia
Number analyzed (Participants) | 10 | 7
Units on a scale | 183.4 (13.86) | 177.2 (16.84)

ADVERSE EVENTS:
Time Frame: To the time the subject was discharged from the hospital.
Description: Hypertension systolic blood pressure greater than 160 mmHg.
Arm/Group | Deep Sedation | General Anesthesia
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/7
Other Adverse Events (participants affected / at risk) | 0/10 | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No